CLINICAL TRIAL: NCT02232334
Title: Effects of Global Osteopathic Manual Treatments on Patients With Idiopathic Gastroparesis
Brief Title: Effects of Global Osteopathic Manual Treatments in Patients With Idiopathic Gastroparesis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Kathleen Brannan Brown, Inc. (Other)
Responsible Party: Principal Investigator, Kathleen Brannan Brown, RN, FNP, CMP DOMP-thesis candidate, Kathleen Brannan Brown, Inc.
Allocation: Non-Randomized | Model: Crossover | Masking: None
Other Study IDs: Brown - 1
Record Dates: First submitted 2014-09-03; First posted 2014-09-05 (Estimated); Last update posted 2015-04-01 (Estimated); Status verified 2015-03

CONDITIONS: Idiopathic Gastroparesis
Keywords: Idiopathic Gastroparesis, Nausea, Vomiting, Abdominal Pain, Gastrectomy, Osteopathy, Gastroparesis Cardinal Symptom Index, GCSI
MeSH Terms: conditions — Nausea; Vomiting; Abdominal Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Osteopathic manual treatment (Experimental): Global Osteopathic Manual treatment: each subject will be treated according to what restrictions or areas of poor mobility are found individually. No two subjects will receive the same overall treatment.
  Interventions: Other: Global Osteopathic Manual Treatment
- Control--no change in current treatment of subject (No Intervention): The population will act as their own control prior to intervention of osteopathy, their will be a control period where the subject maintains current treatment of their gastroparesis. During that period they will fill out the GCSI measuring tool at the beginning of the control period and at the end. Those measurements will be compared to the GSCI results during the intervention period.

INTERVENTIONS:
Other: Global Osteopathic Manual Treatment — subtle manipulations of the body according to the methodology of osteopathic manual therapy will be the intervention on subjects in the study. The global treatments will take into consideration the past medical history of each subject as well as what is found on assessment. Focus is on the position, mobililty and quality of each subjects anatomy.
  Arms: Osteopathic manual treatment

SUMMARY:
Global osteopathic manual treatments will decrease the severity score of the Gastroparesis Cardinal Symptom Index tool of patients with idiopathic gastroparesis.

In this longitudinal controlled pre-test post-test group design, subjects with idiopathic gastroparesis (IG) will be utilized to see if global osteopathic manual treatments can decrease their symptoms. Patients with IG suffer from varying degrees of nausea, vomiting and abdominal pain secondary to delayed gastric emptying. There is no known cause for people suffering from IG.

According to the power analysis, the population will be utilized as the experiment group and the control group. The measuring tool to be used is the Gastroparesis Cardinal Symptom Index (GCSI) which is the most widely used symptom score questionnaire for gastroparesis. The subjects in the population will each fill out the GCSI initially and again after an two (2) week period to measure their symptoms during a control period. The same subjects will then be treated with global osteopathic manual treatments one (1) treatment every two (2) weeks for four (4) weeks (day 1, 14, and 28). The GCSI will be filled out on the day of the first (1st) treatment (which is the last day of the control period) and then two (2) weeks after the last treatment (day 42). In order to reject the null hypothesis, with a p value of < 0.05 and a power of 0.8, a minimum of ten (10) subjects in the treatment group is required with a treatment effect of 1 or more. A 'Treatment effect of 1' is defined by Cohen's d, where d = mean difference/standard deviation.

It is expected that the results will show improvement of symptoms through the data collected from the GCSI questionnaires in the treatment group. The results of this study could be significant and contribute to the osteopathic community validating the effectiveness of traditional osteopathic manual therapy as well as giving non-invasive options to people suffering from the disease since those who struggle with it have minimal treatment options--medicines with significant side effects, full or total stomach removal or gastric electrical stimulator implants.

DETAILED DESCRIPTION:
Gastroparesis is a disorder that presents with delayed gastric emptying, abdominal pain, nausea, and vomiting. This condition can be found in people with complications from diabetes-neuropathy of the vagus nerve and gastric surgery-damage to the vagus nerve. With idiopathic gastroparesis (IG), the cause is poorly understood with theories suggesting viral infections affecting gut motility, pyloric valve spasm as well as damage to the specialized cells within the wall of the stomach. Unfortunately the treatment options are minimal for people suffering from gastroparesis regardless of what type.

It is the action of food propulsion that is poorly understood in regards to IG - specifically smooth muscle, autonomic and enteric nerves and specialized cells in the gut named Interstitial Cells of Cajal (ICC). ICC are the pacemakers cells in the gut that conduct motility.

The objective of this study is to normalize structural abnormalities in patients with idiopathic gastroparesis with global osteopathic manual treatments, using a quantitative research method with a longitudinal controlled pre-test post-test design.

The principal investigator (PI), having a background as an emergency medicine registered nurse, has seen patients in the emergency department suffering from idiopathic gastroparesis. The acute attacks appear intense and debilitating often requiring anti-nausea, pain and anti-anxiety medications. As an osteopathic student, the PI would often wonder what could be achieved with osteopathic manual treatments (OMT) to help these people in the emergency department suffering from these symptoms.

Current treatment available for people suffering from gastroparesis is limited. In his article, Gastroparesis - Current Concepts and Considerations (2008), Dr. Hasler, summarized research and the different treatment options for gastroparesis. There are several medications available for gastroparesis however as discussed by Dr. Hasler, the side effects from these medications are significant.

There are invasive treatments, such as injection of botulinum toxin into the pyloric sphincter, gastric electrical stimulator and gastric resection which have shown some improvement in symptoms but carry heavy risks if utilized.

The research method used to determine if global osteopathic manual treatments can help patients who suffer from idiopathic gastroparesis is a longitudinal pre-test post-test controlled quantitative study. The tool used to measure data is the Gastroparesis Cardinal Index Score (GCSI), which was created by Janssen Global Services, LLC. The GCSI is a reliable and validated tool rating symptom intensity of fullness-early satiety, nausea-vomiting, and bloating. The validation of this tool was tested with 169 subjects who filled out the GCSI and those results were compared with clinician symptom ratings. Total scores of the GCSI were "responsive to changes in overall gastroparesis symptoms as assessed by clinicians (P = 0.0002) and patients (P = 0.002).

A minimum of ten (10) subjects are required for the population according to the power analysis, and at lease twelve (12) subjects will be enrolled to account for the potential 20% drop out rate. However, (20) twenty subjects will be the goal for recruitment for this study. Approval from an Institutional Review Board (IRB) has been acquired through Aspire-IRB, gastroenterologists and family medicine physicians in the Sonoma County and Santa Rosa California area will be given recruitment letters and consent forms with study information to give to patients who qualify for the study. Flyers will be distributed throughout the community (grocery stores, community centers, pharmacies etc.). Social media might be utilized to acquire subjects as there appears to be a strong presence of support groups online of people with gastroparesis.

The entire population, during the control group period, will fill out the GCSI initially and then again at two (2) weeks. Those subjects will transition to the experimental group period of the study-the GCSI filled out on the last day of the control period will be used as the first day of treatment GCSI results. IN the experiment period: the subjects will receive three (3) separate global osteopathic manual treatments over four (4) weeks (day 1, 14, and 28). Two weeks after the third (3rd) treatment (day 42), the subjects will fill out the GCSI a final time. The subjects are waiting two (2) weeks to allow for full integration of the last treatment and the GCSI is designed to record the prior two (2) weeks of patients symptoms.

The subjects in the population will be screened via email and or telephone assuring they meet the inclusion/exclusion criteria. Once consented, each participant will be instructed to fill out the first (1st) GCSI questionnaires and email the completed form back to the PI. The data of the first GCSI completion establishes day one (1) of the two (2) week control period. During the two (2) week control period, subjects are to continue their regular treatments for IG (dietary, medicine). They are not to obtain any new therapies such as massage, acupuncture, osteopathy or start any new conventional medical treatments. If there is an acute attack requiring an emergency room visit, the subject will have to be excluded from the study. At the end of the two (2) week period, those subjects will fill out the GCSI again and those results will be anonymously stored for future data analysis. The subjects then will be transitioned into the experimental period and assigned to have their first treatment. The last day of the control period will start the experimental period. All treatments will occur at the office/clinic of the PI in Santa Rosa California, USA. The PI will be working under her massage practitioner license with malpractice insurance under Associated Bodywork and Massage Professionals (ABMP) as well as Manual Therapy Insurance Plus through the Barral Institute. Both of these institutions cover general and professional liability for massage therapy as well as various forms of manual therapy.

At the first treatment, day one (1) of the experimental period, the GCSI (Appendix A) and health history questionnaire (Appendix I) will have been completed. An anamnesis will be taken and the subject will then be assessed and treated with a global osteopathic manual treatment to treat the lesions found in the assessment. The data from the GCSI will be collected and stored anonymously for data analysis. The lesions found in assessment and techniques used to treat will be stored for use in discussion if appropriate. The process will be repeated at two (2) weeks and four (4) weeks from the first (1st) visit for each participant except without the GCSI and without the health questionnaire as it is only required on the first visit. Each treatment will last ninety (90) minutes. To keep results as consistent as possible, subjects will be seen at the same time of the day for each treatment. The results from two (2) weeks and four (4) weeks will be stored for possible discussion. To allow time for integration of the treatments each participant will fill out the GCSI two (2) weeks after the fourth (4th) week of the experimental period. The data from all GCSI tools filled out from the control and experimental periods will be sent to the PI via email for data analysis.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion criteria for the population is the following: English speaking females or males between the ages of 18-65 with moderate to severe IG--diagnosed by a primary physician or gastro-intestinal physician.

Exclusion Criteria:

* Exclusion criteria for the population: diagnosis of gastroparesis with known cause: secondary to diabetes, post surgical or isolated disorders of motility (Parkinson's disease, non-obstructive pancreatic carcinoma, post-abdominal irradiation, atrophic gastritis, celiac arterial occlusion, Crohn's disease, Chagas disease, varicella zoster), active regular/daily marijuana users or have a diagnosis of cyclical nausea/vomiting abdominal pain secondary to regular marijuana use, alcoholics, history of gastrectomy or current gastric electrical stimulator implant, pregnancy, have any schizoaffective or borderline personality disorder, or received osteopathic manual treatment within the last year.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2014-09; Primary Completion 2015-07 (Estimated); Study Completion 2016-07 (Estimated)

PRIMARY OUTCOMES:
Gastroparesis Cardinal Symptom index | 56 days
  The GCSI is a reliable and validated tool rating symptom intensity of fullness-early satiety, nausea-vomiting, and bloating. The validation of this tool was tested with 169 subjects who filled out the GCSI and those results were compared with clinician symptom ratings. Total scores of the GCSI were "responsive to changes in overall gastroparesis symptoms as assessed by clinicians.

CONTACTS AND LOCATIONS:
Locations (1):
- Kathleen Brannan Brown INC, Santa Rosa, California, United States